CLINICAL TRIAL: NCT02685176
Title: Efficacy of Head and Torso Rewarming by Using a Human Model for Severe Hypothermia
Brief Title: Head and Torso Rewarming Using a Human Model for Severe Hypothermia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2015:101
Record Dates: First submitted 2016-02-12; First posted 2016-02-18 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2018-03

CONDITIONS: Hypothermia
Keywords: hypothermia; rewarming; non-shivering
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No Heat (Experimental): No active heating will be provided post cooling
  Interventions: Other: No heat
- Head (Experimental): Charcoal Heater (STK Heatpac, Emergco Tech Solutions, Vancouver) will be applied to the head following cooling
  Interventions: Device: Charcoal Heater (STK Heatpac, Emergco Tech Solutions, B.C.)
- Torso (Experimental): Charcoal Heater (STK Heatpac, Emergco Tech Solutions, Vancouver) will be applied to the torso following cooling
  Interventions: Device: Charcoal Heater (STK Heatpac, Emergco Tech Solutions, B.C.)

INTERVENTIONS:
Device: Charcoal Heater (STK Heatpac, Emergco Tech Solutions, B.C.) — A heater (STK Heatpac) will be used in the active warming arms of the study.
  Arms: Head; Torso
Other: No heat — No active heating provided post cooling
  Arms: No Heat

SUMMARY:
This Clinical trial is being conducted to study the effectiveness of heat donation through head or torso in hypothermic rewarming efficacy using a human model for severe hypothermia. The purpose of the study is to compare the core rewarming effectiveness of the same amount of heat donation through the head or torso in treatment of hypothermia using a human model for severe hypothermia. The information obtained from this study will give a better understanding of heat-transfer mechanisms. This might help in the ongoing research in hypothermia treatment.

DETAILED DESCRIPTION:
Procedure:

Eight healthy, non-pregnant participants between 18 and 45 years old will be cooled in 8°C water, for 60 minutes or to a core temperature of 35ºC on three occasions and then warmed by each of three warming conditions.

The study will include following specific procedures:

Anthropometric data which includes age, weight, height, and measurements of skinfold thickness at four sites- biceps, triceps, subscapularis, and suprailiac will be collected. Participant's heart rate and electrocardiogram will be monitored continuously throughout the experiment.

Conditions: The three treatment methods are as follows. A. Spontaneous rewarming (Shivering inhibition) In this control condition, Demerol will be infused through the arm or hand vein.

The first 1.5 mg/kg will be slowly injected in five equal doses (of 0.3 mg/kg) at 2 minute intervals during the last 10 minutes of cold water immersion. After removal from the water, further aliquots of 0.3 mg/kg (at minimum of 2-minute intervals) will be given only as necessary to inhibit any shivering that may develop, to a maximum cumulative dose of 3.2 mg/kg body weight.

After towel drying the subject will lie on a mattress under an insulated cover without any extra heating modality. Spontaneous rewarming will be the first condition for every subject, the results will be used to determine the dosage schedule for demerol in the active warming conditions below.

B. Head warming:

Charcoal Heater applied to the Head (CH-H) - A charcoal heater (HEATPAC Personal Heater, Emergco Tech. Solutions, Vancouver) consists of a combustion chamber, a canister containing the charcoal fuel, and a branched heating duct that produces 250 W of heat. The canister is placed inside the combustion chamber and the charcoal fuel is ignited. Heated air is blown through the impermeable heating ducts by a fan within the charcoal heater above the combustion chamber. The combustion chamber will be placed on right side of the face/head with ducts wrapping around the dorsum of the head, anteriorly over the forehead, nose, chin and the neck, not covering the eyes or the mouth. The participant will be breathing ambient air (̴ 22˚C).

C. Torso warming:

Charcoal Heater to the Torso (CH-T) - The same charcoal heater as above will be used. The combustion chamber will be placed on the subject's anterior chest with a towel in between. The flexible ducts will be applied to the areas of high heat transfer i.e. over the shoulders, neck, and then anteriorly under the axillae to cross over the lower anterior chest. Participant will be breathing ambient air at room temperature (~22˚C).

Rewarming procedures will be administered either for a period of 60 minutes or until core temperature returns to normal values ( ̴ 36.5-37˚C). Following that, participants will be placed in a warm water bath (40-42˚C) until they wish to exit or core temperature reaches 37°C.

Research Design:

Each of the three experimental trials will be separated by at least 48 hours. On each of the three trials, participants will be immersed up to the level of the sternal notch in 8˚C for up to 60 minutes or until the core temperature falls to 35˚C. Demerol will be administered by a licensed physician during the final 10 minutes of immersion to suppress shivering. Participants will then exit the water, be dried off and rewarmed with either head or torso warming techniques. After removal from the water, an extra dosage of demerol might be given to suppress shivering only if its necessary. The rewarming will be administered for 120 minutes or until the core temperature returns to normal values (̴36.5-37˚C). The order of warming methods will follow a modified balanced design with control being first and the two active warming conditions being balanced.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults, who answer "No" to all the questions on a Physical Activity Readiness Questionnaire (PAR-Q). Participants will also be interviewed to determine if they have any cardio-respiratory diseases, Raynaud's Syndrome, or any other conditions that can be aggravated by cold exposure.

Exclusion Criteria:

* A positive answer to any PAR-Q question, or any cardio-respiratory diseases, Renal dysfunction, Raynaud's Syndrome, past recreational drug use or any other conditions that can be aggravated by cold exposure.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Rewarming Rate | 120 minutes
  Rate of core temperature increase during rewarming

CONTACTS AND LOCATIONS:
Overall Officials: Gordon G Giesbrecht, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No